CLINICAL TRIAL: NCT00291434
Title: Hyperfractionation and Accelerated Fractionation in Comparison With Conventional Fractionation in Definitive Radiotherapy of Squamous Cell Carcinoma of Larynx, Oropharynx and Hypopharynx
Brief Title: Altered and Conventional Fractionated Radiotherapy in Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Institute of Radiotherapy and Oncology, Macedonia (Other)
Other Study IDs: CF vs HF and AF
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2006-05-04 (Estimated); Status verified 2005-01

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; Fractionation; Radiotherapy; Conventional fractionation; Hyperfractionation; Accelerated fractionation
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The aim of our study was to evaluate the value of two different altered fractionation schedules - hyperfractionation and accelerated fractionation with concomitant boost - in comparison with conventional fractionation in primary definitive radiotherapy for squamous cell carcinomas of the larynx, oropharynx or hypopharynx. The study began and was conducted while the only teletherapy unit in our department was the cobalt-60 machine. During that period we were expecting the installation of new sophisticated equipment. We assumed that the results of this study would be also able to show whether or not it would be rational to use the altered fractionation regimens on the new machines.

DETAILED DESCRIPTION:
Eligible patients admitted from March 1999 to December 2000 were treated with conventionally fractionated radiotherapy. These patients represented the retrospective part of the study. Patients admitted between January 2001 and June 2004 were included in the prospective part of the study. Following the confirmation of their eligibility, altered fractionation schedule assignment was made after stratifying by site of origin (larynx vs oropharynx vs hypopharynx), Karnofsky performance score (60%-70% vs 80%-100%), and stage of disease (I and II vs III and IV). Patients were randomized to receive radiotherapy delivered using either hyperfractionation or accelerated fractionation with concomitant boost as a late accelerating component. Exceptions occurred when patients either refused treatment with two daily fractions or were not offered twice-a-day irradiation because of lack of machine time.

Radiotherapy Scheduling and Technique The conventionally fractionated radiotherapy schedule was 66-70 Gy in 6½ -7 weeks (one fraction of 2 Gy per day, 5 fractions per week), whereas the hyperfractionation treatment schedule was 74.4-79.2 Gy in 6.2-7 weeks (two fractions of 1.2 Gy per day, 10 fractions per week with interfraction interval of at least 6 hours; Figure 1). The treatment schedule in accelerated fractionation using concomitant boost consisted of daily fraction of 1.8 Gy, 5 days a week, up to 32.4 Gy including all sites of disease and electively irradiated areas of the neck, followed by two daily fractions for the last 11-12 days. The first daily fraction encompassed all sites of the disease and electively irradiated neck nodes using a dose of 1.8 Gy, and the second daily fraction was the concomitant boost delivered through reduced fields to encompass the gross disease only, using a fraction of 1.5 Gy up to total doses of 68.7-72 Gy in 6 weeks (Figure 1). The interval between the two daily fractions was at least 6 hours.

ELIGIBILITY:
Inclusion Criteria:The inclusion criteria were age 18-75 years, Karnofsky performance score equal or more then 60%, and all stages of disease except stage IVC (TNM classification according to International Union Against Cancer and American Joint Committee of Cancer (UICC and AJCC) from 1997). -

Exclusion Criteria:Patients with previous or concurrent malignancy other then basal cell carcinoma were excluded.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152
Dates: Start 1999-03; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Valentina B Krstevska, Principal Investigator — 2

REFERENCES:
- [Result] Krstevska V, Crvenkova S. Altered and conventional fractionated radiotherapy in locoregional control and survival of patients with squamous cell carcinoma of the larynx, oropharynx, and hypopharynx. Croat Med J. 2006 Feb;47(1):42-52. PMID 16489696